CLINICAL TRIAL: NCT00177632
Title: Evaluation of Alternative Exercise Treatments on Weight Loss in Overweight Women.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0402119
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-09

CONDITIONS: Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

INTERVENTIONS:
Behavioral: behavioral weight loss

SUMMARY:
The purpose is to examine the additional effect of either yoga or resistance exercise on weight loss weight combined with a standard behavioral weight loss intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. 25-55 years of age
3. BMI = 25-35 kg/m2
4. Ability to provide informed consent.
5. Ability to provide consent from their personal physician to participate in this study.

Exclusion Criteria:

1. Participation in regular exercise (aerobic, yoga or resistance exercise) for > 20 minutes per day on > 2 days per week for the last 3 months. (This study is designed to recruit relatively sedentary adults.)
2. Currently being treated for psychological disorders/conditions and/or currently taking psychotropic medication.
3. Diabetes, hypothyroidism, or other medical conditions which would affect energy metabolism.
4. Women who are currently pregnant, pregnant within the previous six months, or planning on becoming pregnant within the next 12 months. (Pregnancy during initial screening will be based on self-report and will be included on the detailed medical history that is completed by subjects. However, pregnancy status will also be verified by the pregnancy test that is required for the baseline, 6 and 12 month DEXA).
5. Non-medicated resting systolic blood pressure >160 mmHg or non-medicated resting diastolic blood pressure >100 mmHg, or taking medication that would affect blood pressure.
6. Taking medication that would affect resting heart rate or the heart rate response during exercise (e.g., beta blockade).
7. Arrhythmia on resting or exercise electrocardiogram that would indicate that vigorous exercise was contraindicated.
8. History of myocardial infarction or valvular disease.
9. History of orthopedic complications that would prevent optimal participation in the exercise component (e.g., heel spurs, severe arthritis).

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66
Dates: Start 2003-07; Study Completion 2004-07

PRIMARY OUTCOMES:
weight loss

SECONDARY OUTCOMES:
fitness
physical activity
dietary intake
mediators

CONTACTS AND LOCATIONS:
Overall Officials: John M Jakicic, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States